CLINICAL TRIAL: NCT06334640
Title: L'Impatto Del Sonno Nelle Patologie Croniche Oculari
Brief Title: Sleeping Quality and Chronic Ocular Diseases
Acronym: SONNO-OCU
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 37C302
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with glaucoma and macular degeneration: Adults subjects affected by glaucoma and macular degeneration
  Interventions: Diagnostic Test: Three questionaires
- Healthy volunteers: Adult healthy volunteers without eye disease
  Interventions: Diagnostic Test: Three questionaires

INTERVENTIONS:
Diagnostic Test: Three questionaires — Berlin, Pittsburgh and Epworth tests administered during study visit

SUMMARY:
To assess the impact of sleep quality on chronic eyes diseases

DETAILED DESCRIPTION:
In this study 3 questionnaires will be distributed to outpatients attending the routine examinations : the Pittsburgh, the Berlin and the Epworth tests These questionnaires, once completed, will then be collected to be then transformed into digital files for the appropriate statistical evaluations and the drafting of the results and conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with macular degeneration or glaucoma or
* Healthy volunteers

Exclusion Criteria:

- Patients with other ocular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients attending our Institution for scheduled visits/examinations
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of sleep disorders in patients and healthy volunteers | At enrollment
  To analyze the prevalence of sleep disorders in subjects affected by glaucoma and macular degeneration and in healthy volunteers as assessed by Berlin, Pittsburgh and Epworth questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy